CLINICAL TRIAL: NCT00444769
Title: A Multi-Centre, Randomised, Single-Blind, Placebo-Controlled, Parallel Group Study to Investigate the Efficacy of Single Pre-Emptive Doses of GW842166X, a Non-Cannabinoid CB2 Receptor Agonist, on Pain Following Third Molar Tooth Extraction.
Brief Title: Dental Pain 3rd Molar Tooth Extraction GW842166
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBA106809
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Pain
Keywords: analgesia; post-operative pain; GW842166; non-cannabinoid agonist; third molar tooth extraction
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative

INTERVENTIONS:
Drug: GW842166

SUMMARY:
This phase IIa (proof of concept) study will be conducted as a multi-centre study within the European Union (EU). It will be conducted to a randomised, single blind, placebo- controlled, parallel group design with a positive control arm to evaluate the analgesic efficacy of pre-emptive doses of GW842166 following dental surgery (3rd molar tooth extraction). GW842166 will be administered as a single pre-operative oral dose in male and female subjects who will be randomised to take part in one of four possible treatment regimens. Pain assessments will be undertaken over a 10 hr period. Pharmacokinetic blood samples will be collected over a 48 hr period. Safety and tolerability will be evaluated by adverse event monitoring, cardiovascular assessments (ECG and vital signs) and clinical laboratory tests (haematology, clinical chemistry and urinalysis).

ELIGIBILITY:
Inclusion Criteria:

* Body weight = 50 kg and BMI within the range 19 - 29.9 kg/m².
* Women may be of non-child bearing potential or they may be of child-bearing potential. - Women of child-bearing potential must use an effective method of contraception.

Females of non-child bearing potential are defined as:

* Post-menopausal females, being amenorrhoeic for at least 2 years with an appropriate clinical profile, e.g., age appropriate, history of vasomotor symptoms. However, if indicated this should be confirmed by oestradiol and FSH levels consistent with menopause (according to local laboratory ranges).
* Pre-menopausal females with a documented hysterectomy (medical report verification) and/or bilateral oophorectomy. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring and other tests specified in this protocol. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures
* Subject is scheduled for outpatient surgical removal of up to four third molar teeth under local anaesthesia. At least one third molar tooth must be a fully or partially impacted in the mandible requiring bone removal.
* Subject agrees not to take analgesics other than protocol defined rescue analgesics during treatment (up to 48 hrs post dose).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subject has a history or presence of significant organ disease or mental illness.
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody result or positive HIV result within 3 months of screening.
* The subject has a positive pre-study urine drug or urine/breath alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids, Benzodiazepines and Methadone.
* Subject has been exposed to analgesics (including prescription and over the counter NSAIDs or COX-2 inhibitors) within 48 hours or 5 half-lives (whichever is the longer) prior to the start of surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Weighted mean of the pain intensity over the 10 hours post-surgery as measured by the VAS (Visual Analogue Scale) | over the 10 hours post-surgery

SECONDARY OUTCOMES:
-Weighted mean of the pain intensity over the 10 hours post-surgery,measured by the Verbal Rating Scale -VAS and VRS mean pain scores up to 10 hours post-surgery -Elapsed time from study drug administration to rescue analgesic request | over the 10 hours post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, PhD., Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Hamburg, Hamburg, Germany
- GSK Investigational Site, Verona, Veneto, Italy
- GSK Investigational Site, London, United Kingdom